CLINICAL TRIAL: NCT06542601
Title: Effect of Combined Motor and Cognitive Training on Older Adults With Motoric Cognitive Risk Syndrome in Community: a Randomized Controlled Study
Brief Title: Combined Motor and Cognitive Training for Older Adults With Motoric Cognitive Risk Syndrome (CMC-training)
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-234
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-04

CONDITIONS: Disability Physical; Disabilities Mental; Age Problem
Keywords: Motoric Cognitive Risk; Cognitive training; Exercise training

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Total: All subjects
  Interventions: Device: Motor cognitive intervention

INTERVENTIONS:
Device: Motor cognitive intervention — Older adults were given cognitive training and motor training for 12 weeks using a tablet computer

SUMMARY:
To investigate the effects of a combined motor-cognitive intervention on the improvement of motor as well as cognitive function in community residents.

DETAILED DESCRIPTION:
Cognitive training uses systematically designed tasks that are difficulty-adaptive for cognitive domains such as attention, memory, and logical reasoning to improve individual cognitive functioning. Internet-based Adaptive Multi-Cognitive Domain Cognitive Training is conducted 3 times per week for 30 minutes each time, and includes tasks such as delayed memory, paired memory, and inverse numerical breadth.

The exercise intervention was based on the M-Mobile multicomponent exercise program, in which older adults were instructed to complete exercise training at home at least three days per week. In all intervention groups, balance, sitting test and walking speed were assessed according to the Simple Physical Performance Battery (SPPB), and according to their scores, they were given exercise training, including flexibility, balance, aerobic training and resistance training.

ELIGIBILITY:
Inclusion Criteria:

* Age 60-80 years; ≥ 9 years of education; Cognitive impairment: MMSE score 22-26; Slow gait:total walking time >4 seconds and ≤8 seconds in a 4-meter walk test; Agreed to participate in the study and signed an informed consent form.

Exclusion Criteria:

* Dementia/suspected dementia; Suffering from diseases that affect cognitive function, such as cerebrovascular disease, Parkinson's syndrome, etc.; Taking medications related to cognitive improvement and psychiatric disorders, etc.; Recent heart attack, severe cerebrovascular disease, psychiatric disorders, etc.; other inability to persist in completing exercise cognitive interventions, such as suffering from severe musculoskeletal disorders; Participating in another clinical trial at the same time； Participation in an exercise and/or cognitive intervention in the past 6 months; Inability to complete content in studies such as neuropsychological scale assessments.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Study Population: Elderly people with Motoric Cognitive Risk living in Beijing community
Sampling Method: Non-Probability Sample
Enrollment: 204 (Estimated)
Dates: Start 2024-07-04 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive function changes in the intervention group and the control group | 12 weeks
  Changes in Montreal Cognitive Assessment Scale (MoCA) scores before and after intervention between the two groups
Motor function changes in the intervention group and the control group | 12 weeks
  Changes in Montreal Short Physical performance Battery (SPPB) scores before and after intervention between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Yi Tang, MD., PhD., Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China